CLINICAL TRIAL: NCT00624689
Title: Double-blinded Interventional Study on the Effects of MFGM-enriched Formula With Reduced Energy and Protein Content on Growth and Development
Brief Title: Effects of Milk Fat Globule Membrane (MFGM) - Enriched Formula With Reduced Energy and Protein Content on Growth and Development
Acronym: TUMME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Niklas Timby, M.D, Researcher, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TUMME
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Infant
Keywords: Body composition; Glucose tolerance; Intima-media thickness; Visual acuity; Neurological development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Modified formula
  Interventions: Dietary Supplement: Modified formula (MFGM-enriched formula with reduced energy and protein content)
- 2 (No Intervention): Standard formula
- 3 (No Intervention): Breastfed

INTERVENTIONS:
Dietary Supplement: Modified formula (MFGM-enriched formula with reduced energy and protein content) — MFGM-enriched formula with reduced energy and protein content
  Arms: 1

SUMMARY:
Formula-fed infants differ from breast-fed infants in the growth pattern, risk for obesity and cardiovascular diseases, neurological development and morbidity in infections.

The investigators' hypothesis is that a modified formula with reduced energy and protein content and enrichment with Milk Fat Globule Membrane (MFGM) containing bioactive proteins and phospholipids will reduce the difference between formula-fed and breast-fed infants.

ELIGIBILITY:
Inclusion Criteria:

* Term infants with birth weight 2500-4500 gr
* Fed with breastmilk only or formula only before 2 months of age

Exclusion Criteria:

* Chronic illness

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2008-03; Primary Completion 2013-03 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Body composition | 4 months
  Pletysmography (% body fat)

SECONDARY OUTCOMES:
Neurological development | 1 year
  Bayley Scales of Infant and Toddler Development, 3rd Ed (higher score - better outcome)

OTHER OUTCOMES:
Neurological development | 6.5 years
  Wechsler Intelligence Scale for Children, 4th Ed (higher score - better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of clinical sciences, pediatrics, Umeå University, Umeå, Sweden

REFERENCES:
- [Derived] Timby N, Hernell O, Vaarala O, Melin M, Lonnerdal B, Domellof M. Infections in infants fed formula supplemented with bovine milk fat globule membranes. J Pediatr Gastroenterol Nutr. 2015 Mar;60(3):384-9. doi: 10.1097/MPG.0000000000000624. PMID 25714582
- [Derived] Timby N, Domellof E, Hernell O, Lonnerdal B, Domellof M. Neurodevelopment, nutrition, and growth until 12 mo of age in infants fed a low-energy, low-protein formula supplemented with bovine milk fat globule membranes: a randomized controlled trial. Am J Clin Nutr. 2014 Apr;99(4):860-8. doi: 10.3945/ajcn.113.064295. Epub 2014 Feb 5. PMID 24500150